CLINICAL TRIAL: NCT02527291
Title: Cytomegalovirus Reactivation in Non Immunocompromised Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ori Galante, Dr. Ori Galante, Soroka University Medical Center
Other Study IDs: SOR-0231-15-CTIL
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2016-03

CONDITIONS: Cardiac Surgery
Keywords: Cytomegalovirus; Interleukin; Polymerase Chain Reaction; CMV antibodies
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood work: Cytomegalovirus Ab (CMV Ab), Cytomegalovirus Polymerase Chain Reaction (CMV PCR) and Interleukin (IL28).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Study Group: The Study group will comprise of seropositive CMV patients undergoing cardiothorathic surgery and having a complicated postoperative course.
  In addition to the routine blood work which includes: CBC, chemistry and INR, blood work for CMV PCR will be done three times: at enrollment, follow up 1 (7 days post operation) and follow up 2 (14 days post operation).
  Blood work for Interleukin28 (IL28) will be done at enrollment. All visits include data collection from computerized medical records.
  Interventions: Other: Blood test
- Control Group 1: The first control group will be comprised of patients who are seropositive CMV undergoing cardiothorathic surgery and having a normal postoperative course.
  In addition to the routine blood work which includes: CBC, chemistry and INR, blood work for CMV PCR will be done two times: at enrollment and follow up 1 (7 days after discharge).
  Blood work for Interleukin28 (IL28) will be done at enrollment. All visits include data collection from computerized medical records.
  Interventions: Other: Blood test
- Control Group 2: The second control group will include seronegative patients for CMV undergoing cardiothorathic surgery with complicated and uncomplicated post-operative course.
  Blood work for CMV PCR and IL28 will be done at enrollment. All other visits include data collection from computerized medical records only.
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Blood test for CMV PCR and IL28

SUMMARY:
We hypothesized that the stress of cardiac surgery and cardiopulmonary bypass can cause reactivation of a latent CMV infection and that reactivation might be more prevalent in patients with complicated post-operative course. The study aims are:

* To study whether cardiac surgery is a trigger for latent CMV reactivation and to compare reactivation rate between sub groups of patient with complicated post-operative course and non complicated post operative course.
* To study the relationship between expression IL28 SNP rs12979860 and the risk of CMV replication in the non immunocompromised patient undergoing cardiac surgery.

DETAILED DESCRIPTION:
The study population will be screened at the cardiothorathic surgery ward Soroka Medical Center. A member of the study research team will approach individual subjects who are potential candidates (if all inclusion criteria are fulfilled and if there are no exclusion criteria) for participation in the study. The study member will explain the purpose, procedures and intent of the study to each potential participant. Interested patients will be asked to provide written consent prior to performing any study procedure. Each patient will be associated to one group, according to the CMV test results, which will be done at the enrollment.

Study Group - the Study group will comprise of seropositive CMV patients undergoing cardiothorathic surgery and having a complicated postoperative course.

Control Group 1 - the first control group will be comprised of patients who are seropositive CMV undergoing cardiothorathic surgery and having a normal postoperative course.

Control Group 2 - the second control group will include seronegative patients for CMV undergoing cardiothorathic surgery with complicated and uncomplicated post-operative course.

Visit 1 - Screening and enrollment:

After the patient will provide written inform consent data collection will be done by a study member and includes: demographics, clinical and medical information. In addition, vital signs will be taken and blood work: CMV Ab, CMV PCR, CBC, INR, Chemistry and IL28.

Visit 2 - follow up (on the 7th post operative day):

For patients with uncomplicated post operative (post op) course follow up at the cartiothorathic post op clinic one week after discharge. In addition to the routine blood works and medical follow up, a second blood test panel will be drowned including a second CMV PCR for the control group 1. For those patients with complicated post-operative course and prolonged hospitalization a follow up will be done in the cardiothorathic ward and will include medical tracking and blood test for a second CMV PCR for the study group. For control group 2: medical follow up and routine blood works.

Visit 3- follow up 2 (on the 14 th post operative day):

This visit is a follow up for patients still hospitalized post operatively. We will keep medical tracking and draw the last blood test for the 3rd CMV PCR for the study group. For control groups 1 and 2: medical follow up and routine blood works.

Visit 4 - follow up 3 (90 days post op):

Data collection from computerized medical records for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted for cardiac surgery.
2. Age 18 and above.

Exclusion Criteria:

1. Immunosuppressed patients including: HIV, active cancer, biological chemotherapy, steroid use equivalent to prednisone dosage above 1 mg/Kg a day, post organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be screened at the cardiothorathic surgery ward Soroka Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The cumulative of death, prolonged hospitalization, prolonged post-operative mechanical ventilation and prolonged use of vasopressors | 12 months
CMV reactivation: viral load elevation comparing to the baseline level prior to surgery | 12 months

SECONDARY OUTCOMES:
The relationship between expression IL28 SNP rs12979860 and the risk of CMV replication in the non immunocompromised patient undergoing cardiac surgery. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Result] Staras SA, Dollard SC, Radford KW, Flanders WD, Pass RF, Cannon MJ. Seroprevalence of cytomegalovirus infection in the United States, 1988-1994. Clin Infect Dis. 2006 Nov 1;43(9):1143-51. doi: 10.1086/508173. Epub 2006 Oct 2. PMID 17029132
- [Result] Razonable, RR, Limaye, RR. Cytomegalovirus infection after solid organ transplantation. In: Transplant Infections, 3rd ed, Bowden, RA, Ljungman, P, Snydman, DR (Eds), Lippincott Williams and Wilkins, Philadelphia 2010
- [Result] Gavalda, J, Roman, A, Pahissa, A. Risks and epidemiology of infections after lung or heart-lung transplantation. In: Transplant Infections, 3rd edition, Bowden, RA, Ljungman, P, Snydman, DR (Eds), Lippincott Williams and Wilkins, Philadelphia 2010
- [Result] Heininger A, Jahn G, Engel C, Notheisen T, Unertl K, Hamprecht K. Human cytomegalovirus infections in nonimmunosuppressed critically ill patients. Crit Care Med. 2001 Mar;29(3):541-7. doi: 10.1097/00003246-200103000-00012. PMID 11373417
- [Result] Jaber S, Chanques G, Borry J, Souche B, Verdier R, Perrigault PF, Eledjam JJ. Cytomegalovirus infection in critically ill patients: associated factors and consequences. Chest. 2005 Jan;127(1):233-41. doi: 10.1378/chest.127.1.233. PMID 15653989
- [Result] Limaye AP, Kirby KA, Rubenfeld GD, Leisenring WM, Bulger EM, Neff MJ, Gibran NS, Huang ML, Santo Hayes TK, Corey L, Boeckh M. Cytomegalovirus reactivation in critically ill immunocompetent patients. JAMA. 2008 Jul 23;300(4):413-22. doi: 10.1001/jama.300.4.413. PMID 18647984
- [Result] Kalil AC, Florescu DF. Prevalence and mortality associated with cytomegalovirus infection in nonimmunosuppressed patients in the intensive care unit. Crit Care Med. 2009 Aug;37(8):2350-8. doi: 10.1097/CCM.0b013e3181a3aa43. PMID 19531944
- [Result] Wan S, Yim AP, Ng CS, Arifi AA. Systematic organ protection in coronary artery surgery with or without cardiopulmonary bypass. J Card Surg. 2002 Nov-Dec;17(6):529-35. doi: 10.1046/j.1540-8191.2002.01010.x. PMID 12643464
- [Result] Booth D, George J. Loss of function of the new interferon IFN-lambda4 may confer protection from hepatitis C. Nat Genet. 2013 Feb;45(2):119-20. doi: 10.1038/ng.2537. PMID 23358218
- [Result] Kelly C, Klenerman P, Barnes E. Interferon lambdas: the next cytokine storm. Gut. 2011 Sep;60(9):1284-93. doi: 10.1136/gut.2010.222976. Epub 2011 Feb 8. PMID 21303914
- [Result] Rauch A, Kutalik Z, Descombes P, Cai T, Di Iulio J, Mueller T, Bochud M, Battegay M, Bernasconi E, Borovicka J, Colombo S, Cerny A, Dufour JF, Furrer H, Gunthard HF, Heim M, Hirschel B, Malinverni R, Moradpour D, Mullhaupt B, Witteck A, Beckmann JS, Berg T, Bergmann S, Negro F, Telenti A, Bochud PY; Swiss Hepatitis C Cohort Study; Swiss HIV Cohort Study. Genetic variation in IL28B is associated with chronic hepatitis C and treatment failure: a genome-wide association study. Gastroenterology. 2010 Apr;138(4):1338-45, 1345.e1-7. doi: 10.1053/j.gastro.2009.12.056. Epub 2010 Jan 11. PMID 20060832
- [Result] Tanaka Y, Nishida N, Sugiyama M, Kurosaki M, Matsuura K, Sakamoto N, Nakagawa M, Korenaga M, Hino K, Hige S, Ito Y, Mita E, Tanaka E, Mochida S, Murawaki Y, Honda M, Sakai A, Hiasa Y, Nishiguchi S, Koike A, Sakaida I, Imamura M, Ito K, Yano K, Masaki N, Sugauchi F, Izumi N, Tokunaga K, Mizokami M. Genome-wide association of IL28B with response to pegylated interferon-alpha and ribavirin therapy for chronic hepatitis C. Nat Genet. 2009 Oct;41(10):1105-9. doi: 10.1038/ng.449. Epub 2009 Sep 13. PMID 19749757
- [Result] Egli A, Levin A, Santer DM, Joyce M, O'Shea D, Thomas BS, Lisboa LF, Barakat K, Bhat R, Fischer KP, Houghton M, Tyrrell DL, Kumar D, Humar A. Immunomodulatory Function of Interleukin 28B during primary infection with cytomegalovirus. J Infect Dis. 2014 Sep 1;210(5):717-27. doi: 10.1093/infdis/jiu144. Epub 2014 Mar 11. PMID 24620020
- [Result] Bravo D, Solano C, Gimenez E, Remigia MJ, Corrales I, Amat P, Navarro D. Effect of the IL28B Rs12979860 C/T polymorphism on the incidence and features of active cytomegalovirus infection in allogeneic stem cell transplant patients. J Med Virol. 2014 May;86(5):838-44. doi: 10.1002/jmv.23865. Epub 2013 Dec 27. PMID 24374819